CLINICAL TRIAL: NCT06727409
Title: Use of Clinical-trials and Simulation Models to Estimate Cost-effectiveness of Non-steroidal Mineralocorticoid Antagonists, RASi and SGLT2i as Triple Therapy With Type 2 Diabetes and Chronic Kidney Disease
Acronym: RAiSiN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Elaine Chow, Clinical Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAiSiN; CREC number: 2023.615-T (Other: CUHK Clinical Research Ethics Committee)
Record Dates: First submitted 2024-11-29; First posted 2024-12-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-12

CONDITIONS: Patients With Type 2 Diabetes
Keywords: Finereone, Triple therapy, Type 2 Diabetes, Chronic kidney disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — finerenone

STUDY DESIGN:
Intervention Model Description: in parallel fashion to optimise tolerated doses of Finerenone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Finerenone on top of maximal tolerated RASi and stable SGLT2i therapy (Experimental): pre and post Finerenone treatment evaluation
  Interventions: Drug: Finerenone

INTERVENTIONS:
Drug: Finerenone — Finerenone 10mg or 20 mg as tolerated on top of maximal tolerated RASi and stable SGLT2i therapy

SUMMARY:
To evaluate triple therapy with nsMRA, RASi and SGLT2i on albuminuria in individuals with T2D and CKD

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above
* Diagnosis of type 2 diabetes at least 6 months
* CKD (eGFR by CKD-EPI 25-90 ml/min/1.73m2 with uACR 30 to <300 mg/g) and/or those with severely elevated albuminuria (uACR 30-5000 mg/g) and eGFR > 60 ml/min/1.73m2.
* Patients should have a serum potassium <4.8 mmol/l at screening
* On SGLT2i (dapagliflozin or empaglifozin) at screening at stable doses for at least 4 weeks.
* On ACEi or ARB at maximum tolerated dose per manufacturer's label that did not cause unacceptable side effects
* In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a suitable study candidate.

Exclusion Criteria:

* Type 1 diabetes
* Allergy, contraindications or intolerance to ACEi/ARB
* Contraindications or intolerance to mineralocorticoid receptor antagonists
* Allergy, contraindications to SGLT2is
* Currently pregnant or planning pregnancy
* HbA1c >9% at enrolment
* Uncontrolled hypertension SBP > 160mmHg or hypotension <90 mmHg at enrolment
* Concomitant therapy with eplenerone, spironolactone that cannot be discontinued.
* History of stroke or worsening heart failure in the past 6 months prior to screening
* Diabetic ketoacidosis, hyperosmolar hyperglycaemic state or myocardial infarction in the six months prior to screening
* Patients on renal replacement therapy or likely require kidney transplant or dialysis during the study period
* On concomitant strong CYP3A4 inhibitors that cannot be discontinued
* Adrenal insufficiency
* Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
* An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in urine albumin creatinine ratio (uACR) | 26 weeks
  urine ACR between baseline and end of study (26 weeks)

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) | 26 weeks
  eGFR calculated from plasma creatinine from baseline to end of study in ml/min/1.73m2
Change in potassium | 26 weeks
  Change in plasma potassium (mmol/l) from baseline to end of study
Change in blood pressure | 26 weeks
  Change in systolic and diastolic blood pressure (mmHg) from baseline to end of study
Change in heath related quality of life | 26 weeks
  change in HRQoL from baseline to end of study using EQ5D
Change in body weight | 26 weeks
  Change in body weight (kg) from baseline to end of study

CONTACTS AND LOCATIONS:
Locations (1):
- 3M, Diabetes and Endocrine Research Center, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes